CLINICAL TRIAL: NCT02994680
Title: Effects of a Liquefied Petroleum Gas Stove and Fuel Distribution Intervention on Adult Cardiopulmonary Health Outcomes in Puno, Peru
Brief Title: Cardiopulmonary Outcomes and Household Air Pollution Trial
Acronym: CHAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Washington University School of Medicine (Other); University of Georgia (Other); Emory University (Other); Universidad Peruana Cayetano Heredia (Other); Asociacion Benefica Prisma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00007128
Record Dates: First submitted 2016-11-28; First posted 2016-12-16 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2020-07

CONDITIONS: Blood Pressure; Carotid Intima Media Thickness; Endothelial Function; Signs and Symptoms, Respiratory; Respiratory Function Tests
Keywords: Air Pollution; Liquefied Petroleum Gas; Cookstove; Behavioral Intervention; Propane Stove
MeSH Terms: conditions — Signs and Symptoms, Respiratory

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: The clinical team is masked in this study, and a portion of the investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Will receive:
  1. Three-burner LPG stove (at enrollment)
  2. Delivery of LPG tanks (beginning at enrollment for one year)
  The study will be conducted over three years, with staggered enrollment over one year, one year of observations during the intervention period, and one year of follow-up observations after the intervention period for each participant.
  Participants in the intervention arm will receive an LPG stove upon enrollment and the research team will deliver fuel twice monthly to their homes during the first year. Participants in the intervention arm will not receive fuel during the second year, but researchers will encourage these participants to continue using LPG fuel for cooking.
  Interventions: Device: Three-burner LPG stove; Other: Delivery of LPG tanks
- Control arm (Active Comparator): Will receive:
  1. Three-burner LPG stove (one year after enrollment)
  2. Vouchers for LPG tanks (one year after enrollment)
  Participants in the control arm but will not receive an LPG stove or fuel during the first year. Instead, participants will receive an LPG stove at the end of the first year and vouchers to obtain free fuel at distribution centers during the course of the second year.
  Interventions: Device: Three-burner LPG stove; Other: Vouchers for LPG tanks

INTERVENTIONS:
Device: Three-burner LPG stove — The intervention arm will receive a three-burner LPG stove upon enrollment. The control arm will receive the stove one year after enrollment.
  Other Names: propane stove; SURGE three-burner liquefied petroleum gas stove
Other: Delivery of LPG tanks — One year supply of LPG fuel, in the form of delivery of 20 kg tank that holds 10 kg of LPG. Delivered to homes.
  Other Names: propane tank
  Arms: Intervention arm
Other: Vouchers for LPG tanks — One year supply of LPG, in the form of vouchers to obtain a free LPG tanks from a distribution center. (Beginning one year after enrollment, for one year)
  Other Names: coupon
  Arms: Control arm

SUMMARY:
The purpose of this randomized controlled field trial is to determine whether a liquefied petroleum gas (LPG) stove and fuel distribution intervention reduces personal and kitchen exposure to household air pollutants and improves cardiopulmonary health outcomes when compared to usual cooking practices with open-fire biomass-burning stoves in adult women aged 25-64 years.

DETAILED DESCRIPTION:
Randomized, controlled field trial of an LPG stove and fuel distribution intervention compared to standard cooking practices with open-fire biomass-burning stoves in the homes of participating adult women aged 25-64 years. The aim is to determine whether provision of cleaner fuels will result in important reductions in household air pollutants and consequently in an improvement in cardiopulmonary health outcomes over a one-year period. Participants randomly assigned to the intervention arm will receive a free LPG stove and fuel delivered to their homes during the one-year intervention period. Participants randomly assigned to the control arm will receive a free LPG stove and vouchers that can be used to obtain free fuel for an entire year at LPG fuel distribution centers at the end of the one-year intervention period. All participants will be followed for a second year to assess patterns and impacts of sustained use (intervention arm) and initial adoption (control arm).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Full-time resident ≥6 months in current location
* Capable of understanding procedures
* Capable of providing informed consent and responding to a questionnaire
* Primary household cook
* Currently using a traditional stove as primary stove for cooking
* Cooking room/area separate from sleeping room/area to minimize probability of use of biomass fuel stoves for heating living space.

Exclusion Criteria:

* Plans to move from the area within one year
* Uncontrolled hypertension
* Diagnosis of chronic obstructive pulmonary disease (COPD)
* Pregnant or planning pregnancy in the next year

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Particulate matter of 2.5 μm in size (household air pollutant) | One year
  Specific Aim: Demonstrate sustained reductions in personal and kitchen particulate matter concentrations after distribution of an LPG stove and fuel tanks twice monthly over a one-year period.
  Hypothesis: Use of LPG stoves for cooking by participants in the intervention arm will result in a sustained reduction in personal and kitchen air pollutant concentrations when compared to those with the control arm during the one year intervention period.
Carbon monoxide (household air pollutant) | One year
  Specific Aim: Demonstrate sustained reductions in personal and kitchen carbon monoxide concentrations after distribution of an LPG stove and fuel tanks twice monthly over a one-year period.
  Hypothesis: Use of LPG stoves for cooking by participants in the intervention arm will result in a sustained reduction in personal and kitchen carbon monoxide concentrations when compared to those with the control arm during the one year intervention period.
Blood pressure (cardiovascular health endpoint) | One year
  Specific Aim: Demonstrate sustained reduction in blood pressure after LPG stove intervention.
  Hypothesis: Women in the intervention arm will have lower blood pressure when compared with those in the control arm during the one year intervention period.
Flow mediated dilation (cardiovascular health endpoint) | One year
  Specific Aim: Demonstrate a sustained improvement in endothelial function after LPG stove intervention.
  Hypothesis: Women in the intervention arm will have better endothelial function as measured by flow mediated dilation when compared with those in the control arm during the one year intervention period.
Carotid intima media thickness (cardiovascular health endpoint) | One year
  Specific Aim: Demonstrate lower progression in carotid intima media thickness after LPG stove intervention.
  Hypothesis: Women in the intervention arm will have a lower rate of atherosclerosis progression as measured by carotid artery ultrasound assessment of the carotid intima-media complex over a one-year period when compared with those in the control arm during the one year intervention period.
Respiratory symptoms (respiratory health endpoint) | One year
  Specific Aim: Demonstrate sustained reduction in respiratory symptoms after LPG stove intervention.
  Hypothesis: Women in the intervention arm will have fewer respiratory symptoms as measured by a lower St. Georges Respiratory Symptoms Questionnaire score when compared with those in the control arm during the one year intervention period.
Peak expiratory flow (respiratory health endpoint) | One year
  Specific Aim: Demonstrate sustained improvement in peak expiratory flow after LPG stove intervention.
  Hypothesis: Women in the intervention arm will have a higher peak expiratory flow as measured by spirometry when compared with those in the control arm during the one year intervention period.
Forced expiratory volume at one second (respiratory health endpoint) | One year
  Specific Aim: Demonstrate higher forced expiratory volumes at one second after LPG stove intervention.
  Hypothesis: Women in the intervention arm will have higher height- and age-adjusted, pre- and post-bronchodilator forced expiratory volume at one second as measured by spirometry over a one-year period when compared with those in the control arm during the one year intervention period.

SECONDARY OUTCOMES:
Quality-adjusted life years | One year
  Specific Aim: Demonstrate improvements in quality of life scores after LPG stove intervention, as calculated by the Short Form-36 questionnaire.
  Hypothesis: Women in the intervention arm will have better quality of life related score than those in the control arm at the end of the one year intervention period.
Inflammatory metabolites | One year
  Specific Aim: Demonstrate reductions in inflammatory metabolites measured in urine and dot blood samples after LPG stove intervention.
  Hypothesis: Women in the intervention arm will have lower concentrations of inflammatory metabolites in urine and dot blood samples when compared to those in the control arm during the one year intervention period.
Compliance with stove use | One year
  Hypothesis: Stove use monitors will demonstrate >90% compliance with LPG stove use during the one-year intervention period in the LPG stoves of participants in the intervention arm.
Exhaled carbon monoxide | One year
  Specific Aim: Demonstrate sustained lower exhaled carbon monoxide concentrations during the one-year intervention period.
  Hypothesis: Personal exhaled carbon monoxide concentrations will be lower in participants in the intervention arm when compared to those in the control arm.
Diet | One year
  Specific Aim: Document changes in diet after LPG stove intervention, as measured by 24-hour recalls.
  Hypothesis: Women in the intervention arm will have a better diet than those in the control arm during the one year intervention period.
Urinary sodium | One year
  Specific Aim: Document changes in salt intake after LPG stove intervention, as measured by 24-hour recalls.
  Hypothesis: Women in the intervention arm will have lower urinary sodium than those in the control arm after the intervention.
Percentage of households with sustained LPG stove use in intervention arm | One year
  Hypothesis: Participants in the intervention arm will continue to use their LPG stoves without stove stacking in the year following the intervention.
Percentage of households who adopted LPG stove use in the control arm | One year
  Specific Aim: Characterize the percentage of participants in control arm who decided to adopt LPG stove use one year after the intervention.
  Hypothesis: Participants in the control arm will adopt LPG stoves without stove stacking in the year following the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: William N Checkley, MD, PhD, Principal Investigator — Associate Professor
Locations (1):
- Puno Global Non-Communicable Disease Research Site, School of Medicine, Johns Hopkins University, Puno, Peru

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual patient data (IPD).

REFERENCES:
- [Background] Fandino-Del-Rio M, Goodman D, Kephart JL, Miele CH, Williams KN, Moazzami M, Fung EC, Koehler K, Davila-Roman VG, Lee KA, Nangia S, Harvey SA, Steenland K, Gonzales GF, Checkley W; Cardiopulmonary outcomes and Household Air Pollution trial (CHAP) Trial Investigators. Effects of a liquefied petroleum gas stove intervention on pollutant exposure and adult cardiopulmonary outcomes (CHAP): study protocol for a randomized controlled trial. Trials. 2017 Nov 3;18(1):518. doi: 10.1186/s13063-017-2179-x. PMID 29100550
- [Derived] Fandino-Del-Rio M, Kephart JL, Williams KN, Shade T, Adekunle T, Steenland K, Naeher LP, Moulton LH, Gonzales GF, Chiang M, Hossen S, Chartier RT, Koehler K, Checkley W; Cardiopulmonary outcomes and Household Air Pollution (CHAP) Trial Investigators. Household Air Pollution Concentrations after Liquefied Petroleum Gas Interventions in Rural Peru: Findings from a One-Year Randomized Controlled Trial Followed by a One-Year Pragmatic Crossover Trial. Environ Health Perspect. 2022 May;130(5):57007. doi: 10.1289/EHP10054. Epub 2022 May 12. PMID 35549716
- [Derived] Checkley W, Williams KN, Kephart JL, Fandino-Del-Rio M, Steenland NK, Gonzales GF, Naeher LP, Harvey SA, Moulton LH, Davila-Roman VG, Goodman D, Tarazona-Meza C, Miele CH, Simkovich S, Chiang M, Chartier RT, Koehler K; CHAP Trial Investigators. Effects of a Household Air Pollution Intervention with Liquefied Petroleum Gas on Cardiopulmonary Outcomes in Peru. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2021 Jun 1;203(11):1386-1397. doi: 10.1164/rccm.202006-2319OC. PMID 33306939